CLINICAL TRIAL: NCT05224713
Title: Correlations Between Press Ganey Hospital and Ambulatory Scores for a Neurosurgical Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 015.MBSI.2021.A
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a retrospective review of MHS neurosurgeon hospital (i.e., Methodist Dallas Medical Center, Methodist Richardson Medical Center, Methodist Charlton Medical Center, and Methodist Mansfield Medical Center) and ambulatory clinics (Methodist Moody Brain and Spine Institute [MBSI]- Dallas, MBSI-Richardson, MBSI-Mansfield, MBSI-Sunnyvale, MBSI-Charlton, MBSI-Grand Prairie, and MBSI-Park Cities) PG HCAHPS survey results received between January 1, 2016 and December 31, 2020.

DETAILED DESCRIPTION:
This will be a retrospective review of MHS neurosurgeon hospital (i.e., Methodist Dallas Medical Center, Methodist Richardson Medical Center, Methodist Charlton Medical Center, and Methodist Mansfield Medical Center) and ambulatory clinics (Methodist Moody Brain and Spine Institute [MBSI]- Dallas, MBSI-Richardson, MBSI-Mansfield, MBSI-Sunnyvale, MBSI-Charlton, MBSI-Grand Prairie, and MBSI-Park Cities) PG HCAHPS survey results received between January 1, 2016 and December 31, 2020. Patient electronic medical records will also be reviewed to identify details including: demographics, and chief complaints or indication, and/or procedure details. We anticipate completing this review by September 2021

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Completed a PG HCAHPS hospital and/or ambulatory survey between January 1, 2016 and December 31, 2020 in relation to a MHS neurosurgeon hospital and/or ambulatory visit

Exclusion Criteria:

• Patients not meeting the study inclusion criteria in section 4.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age 18 years or older
  * Completed a PG HCAHPS hospital and/or ambulatory survey between January 1, 2016 and December 31, 2020 in relation to a MHS neurosurgeon hospital and/or ambulatory visit
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-07-06 (Estimated); Study Completion 2024-07-06 (Estimated)

PRIMARY OUTCOMES:
Care provider (CP) overall - section score of CP domains | June 2021 - September 2021
  includes: friendliness/courtesy of CP; CP explanations of problems/condition; CP concern for questions/worries; CP efforts to include in decisions; CP information about medications; CP instructions for follow-up care; CP spoke using clear language; time CP spent with patient; patients' confidence in CP; and likelihood of recommending CP.
Likelihood to recommend CP to others | June 2021 - September 2021
  (Single question)
Overall - Mean survey score of all PG ambulatory survey sections | June 2021 - September 2021
  access overall; billing overall; nurse/assistant overall; CP overall; personal issues overall; and assessment of care overall
Doctors overall - section score of care provider domain | June 2021 - September 2021
  includes: time physician spent with you; physician's concern for your questions and worries; and how well physician kept you informed
Likelihood of recommending hospital to others | June 2021 - September 2021
  (single question)
Overall rating of care given at hospital | June 2021 - September 2021
  (single question)
Overall - mean survey score of all PG hospital survey sections | June 2021 - September 2021
  includes: personal issue overall; nurses overall; overall assessment; doctors overall; and room overall

SECONDARY OUTCOMES:
Trends in PG mean score for each survey question, each section, and overall, by year and by de-identified surgeon | June 2021 - September 2021
  Trends in PG mean score for each survey question, each section, and overall, by year and by de-identified surgeon
Differences by patient demographics | June 2021 - September 2021
  Differences by patient demographics

CONTACTS AND LOCATIONS:
Overall Officials: Richard Meyrat, MD, Principal Investigator — Methodist
Locations (1):
- Methodist Moody Brain and Spine Institute, Methodist Dallas Medical Center, Dallas, Texas, United States